CLINICAL TRIAL: NCT07064811
Title: Standardized Resistance Training Program and Assessment System for Prostate Cancer Patients Receiving Androgen Deprivation Therapy ISPoRT-PCa-ADT Study Protocol for a Randomized Controlled Trial. SPORT-MU
Acronym: SPORT-MU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPORT-MU
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPORT Protocol intervention (Experimental): 24 week velocity based resistance training. Twice weekly supervised sessions
  Interventions: Procedure: SPoRT-Control Intervention
- SPORT Control intervention (Active Comparator): 24-week home based resistance training program .
  Interventions: Procedure: Exercise Intervention Protocol

INTERVENTIONS:
Procedure: Exercise Intervention Protocol — Subjects participated in the supervised exercise program twice weekly (with a 48-72-hour interval between sessions) for 24 weeks, totaling 48 supervised sessions. The progressive resistance training program used velocity-based training principles [24-26], a novel approach in exercise oncology that allows for precise load management and indi-vidualization based on daily performance capacity
  Arms: SPORT Control intervention
Procedure: SPoRT-Control Intervention — structured written instructions for a personalized home-based resistance training program. The protocol was designed to prioritize safety, progressive adaptation, and individualization based on each participant's functional capacity and available resources at home. The program was intended to be performed two to three times per week on non-consecutive days, focusing exclusively on lower-body training through a single primary movement. Each session consisted of three effective sets of 12 repetitions, which served as the standard training volume for the main exercise.
  Arms: SPORT Protocol intervention

SUMMARY:
This randomized controlled trial (RCT) with two parallel study arms evaluated the effectiveness of a 24-week exercise intervention in prostate cancer (PCa) patients under-going androgen deprivation therapy (ADT). Ethical approval was obtained from the Clinical Research Ethics Committee of the University Clinical Hospital "Virgen de la Arrixaca" (Murcia, Spain). Participants were randomly assigned to one of two groups: (1) a supervised progressive resistance training program (SPoRT-PCa-ADT), or (2) a control group receiving a home-based exercise protocol following an initial assessment, accom-panied by weekly telephone follow-up. Assessments were conducted at baseline and at 24 weeks to examine changes in physical, functional, and psychosocial outcomes. Addi-tionally, patient-reported outcomes were collected at the 12-week midpoint (Figure 1). This study design enabled the evaluation of both immediate and sustained intervention effects and facilitated a direct comparison between supervised and home-based exercise approaches

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) with two parallel study arms evaluated the effectiveness of a 24-week exercise intervention in prostate cancer (PCa) patients under-going androgen deprivation therapy (ADT). Ethical approval was obtained from the Clinical Research Ethics Committee of the University Clinical Hospital "Virgen de la Arrixaca" (Murcia, Spain). Participants were randomly assigned to one of two groups: (1) a supervised progressive resistance training program (SPoRT-PCa-ADT), or (2) a control group receiving a home-based exercise protocol following an initial assessment, accom-panied by weekly telephone follow-up. Assessments were conducted at baseline and at 24 weeks to examine changes in physical, functional, and psychosocial outcomes. Addi-tionally, patient-reported outcomes were collected at the 12-week midpoint (Figure 1). This study design enabled the evaluation of both immediate and sustained intervention effects and facilitated a direct comparison between supervised and home-based exercise approaches

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of locally advanced or metastatic prostate neoplasm and current treatment with androgen deprivation therapy (ADT)
* treatment at the radiotherapy oncology department of University Clinical Hospital "Virgen de la Arrixaca"
* legal adult age with signed informed consent

Exclusion Criteria:

* unwillingness to participate in the study
* inability to complete adequate follow-up due to any cause that would prevent knowledge of patient evolution during the follow-up period
* no controlled or symptomatic metastatic bone disease
* physical disabilities that would prevent participants from safely completing the exercise protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate
Enrollment: 60 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Progressive loading test | Up for a 24 weeks
  squat (SQ) exercise to evaluate strength and velocity parameters. Participants performed the SQ starting from an upright position with knees and hips fully extended, feet parallel and shoulder-width apart, and the bar resting on the upper back at the acromion level. Each participant descended continuously until the top of the thighs were below the horizontal plane, with the posterior thighs and shins in contact (~35-40° knee flexion), then immediately reversed the movement to return to the upright position.
Vertical jump test | up for 24 weeks
  In the countermovement jump (CMJ) test, participants performed five maximum CMJs with 20-second rests between jumps. Before CMJ evaluation, participants warmed up by performing two sets of 10 squats without external load, 5 submaximal CMJs, and 3 maximum CMJs. CMJ height was calculated from flight time values determined using a contact platform (Chronojump Boscosystem®, Barcelona, Spain). After discarding the highest and lowest CMJ heights, the resulting average was retained for further analysis. This test was employed as a measure of lower body power and neuromuscular function, which are commonly impaired in patients undergoing ADT.
Maximum Isometric Contraction Test | up for 24 weeks
  Maximum isometric force (MIF) and maximum rate of force development (RFDmax) were measured during a maximum voluntary isometric contraction (MVIC) test in the squat (SQ) exercise with participants standing and knees flexed at 90° (180° = full exten-sion). This test was performed on a quadriceps extension machine. Participants were in-structed to push against the force platform as quickly and forcefully as possible following the "ready, set, go!" signal during two 5-second trials separated by 1-minute rests. External forces were recorded at a sampling rate of 1000 Hz and processed using specific software (Chronojump Boscosystem®, Barcelona, Spain). RFDmax was calculated as the maximum slope in the time-force curve over 20 ms intervals. Additionally, the average tangential slope of the time-force curve obtained at different time intervals (50, 100, and 150 ms from the onset of force production, RFD0-50, RFD0-100, and RFD0-150, respec-tively) was calculated. The average value of each var
Fatigue assessment | Up for 24 weeks
  Cancer-related fatigue, one of the most common and debilitating side effects of cancer treatment and ADT, was assessed using the Brief Fatigue Inventory (BFI). This validated 9-item questionnaire measures the severity of fatigue and its interference with daily activities. Scores are categorized as mild (1-3), moderate (4-6), or severe (7-10) fatigue. The BFI has demonstrated excellent reliability and validity in cancer populations and is sensitive to changes following exercise interventions
Quality of Life Assessment | Up for a 24 weeks
  Quality of life was evaluated using the Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire. This 39-item instrument comprises the FACT-General (FACT-G) plus a prostate cancer subscale (PCS) that assesses concerns specific to prostate cancer and its treatment. The FACT-P evaluates physical wellbeing, social/family wellbeing, emotional wellbeing, functional wellbeing, and prostate cancer-specific concerns. Higher scores indicate better quality of life. This instrument has been extensively validated in prostate cancer populations and demonstrates good sensitivity to change following interventions
Psychological Distress | Up for 24 weeks
  Psychological distress was assessed using the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire designed to identify anxiety and depression in patients with physical health problems. The scale produces separate scores for anxiety and depression. The HADS has been validated in cancer populations and is widely used in psycho-oncology research
Urinary Function | Up for a 24 weeks
  Urinary function, which can be affected by both prostate cancer and its treatments, was assessed using the International Prostate Symptom Score (IPSS). This 8-item questionnaire evaluates the severity of lower urinary tract symptoms associated with benign prostatic hyperplasia and other conditions affecting urinary function in men. The total symptom score ranges from 0 to 35, with higher scores indicating more severe symptoms. Additionally, includes an ancillary query regarding the patient's quality of life related to urinary symptoms, thereby providing a comprehensive evaluation that supports both diagnostic and therapeutic decision-making in clinical practice
Sleep Quality | Up for a 24 weeks
  Sleep disturbances are common in cancer patients and can significantly impact quality of life. Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-report questionnaire that evaluates sleep quality and disturbances over a one-month period

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Soler López, Principal Investigator — Department of Physical Activity and Sport, Faculty of Sport Science, University of Murcia,
Locations (1):
- HCUVA, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided